CLINICAL TRIAL: NCT05196009
Title: Breaking Systems Barriers for Trans Women of Color Living With HIV
Brief Title: mHealth Systems Navigation- Breaking Systems Barriers for Trans Women Living With HIV
Acronym: mSN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-34978
Record Dates: First submitted 2021-11-15; First posted 2022-01-19 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-02

CONDITIONS: Mental Health Issue; Substance Use
Keywords: HIV; Transgender Women; Implementation Science
MeSH Terms: conditions — Substance-Related Disorders | interventions — Mental Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental Health and Substance Use support (Experimental): Pilot Mental health and substance use peer navigation, ecological momentary assessments and virtual support group
  Interventions: Behavioral: mHealth peer navigation and social support

INTERVENTIONS:
Behavioral: mHealth peer navigation and social support — Peer navigation, asynchronous support via SMS, Motivational Interviewing, virtual social support group focused on mental health and substance use, linkage and follow-up
  Other Names: Mental Health and Substance use linkage and initiation support

SUMMARY:
The proposed study will test a mHealth peer navigation intervention for trans women living with HIV in a trans public health clinics to increase initiation and engagement in mental health and substance use services. The peer will navigate and provide support in-person and via mobile phone with HIPAA-compliant text messaging. Ecological momentary assessments will be conducted to enhance self-monitoring of mental health stress and coping-related substance use.

DETAILED DESCRIPTION:
Trans women carry the largest population burden of HIV in San Francisco and have low utilization of mental health and substance use services. The investigators' goal is to use lessons learned in a prior previously-funded Special Projects of National Significance to conduct a pilot peer delivered mHealth support and navigation intervention for trans women living with HIV. The investigators will work with partners in San Francisco Department of Public Health (SFDPH) clinics. The SFDPH is a HRSA-funded entity with trans-specific clinics and a host of in-house referrals to trans-competent mental health and substance use services. Despite availability of trans-specific services, considerable systems barriers exist. Trans clinics have limited clinic hours, and providers have large patient loads wherein medical gender affirmation and HIV care needs must be attended to in short visits. Visit and clinic time and large patient volume leaves providers with little time to ensure continuity in mental health and substance use referrals. To overcome these issues, a peer navigator will deliver mobile and in-person support and navigation to increase substance use and mental health service initiation and engagement among trans women living with HIV in trans health clinics. The research team has already conducted formative research with community members, key stakeholders and providers in San Francisco to help shape and refine the intervention model during the implementation phase of the research.In the implementation phase, the research team will pilot the mSN intervention to improve initiation and engagement in mental health and substance use (MHSU) services.

ELIGIBILITY:
Inclusion Criteria:

* Intervention study:

  1. Provision of signed and dated informed consent form
  2. Declaration of willingness to comply with all study procedures and availability during the study
  3. Age 18 years old or older
  4. Male sex designated at birth
  5. Identify as trans woman, woman or another gender identity not associated with being a man
  6. Desire to join the mSN intervention
  7. Access to a cell phone compatible with social networks (smartphone) to participate in a technology-based intervention or willing to use a study provided cell phone
  8. Speaks English or Spanish
  9. Living in San Francisco Bay Area
  10. Attend a clinic within the San Francisco Department of Public Health

Potential participants living with HIV must meet the following criteria:

1. Documented diagnosis of HIV infection
2. Have missed one recent HIV care appointment or have a detectable viral load
3. Have not initiated or are regularly engaged in mental health and/or substance use services
4. Screen positive for having an alcohol disorder OR drug misuse OR screen positive for psychological distress.

Exclusion Criteria:

1. Participation in another intervention study to promote HIV care in the last year or participation in another study that prevents concomitant inclusion (co-enrollment)
2. Any health condition that, in the investigator's opinion, makes it impossible to participate in the study or impairs the potential participant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans women
Enrollment: 40 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Mental health services initiation | 12 months
  The proportion of participants enrolled in the study who initiate mental health services.
Substance use services initiation | 12 months
  The proportion of participants enrolled in the study who initiate substance use services.
Mental health services engagement | 12 months
  The proportion of participants who remain enrolled in mental health services throughout the follow-up period.
Substance use services engagement | 12 months
  The proportion of participants who remain enrolled in substance use services throughout the follow-up period.

SECONDARY OUTCOMES:
Patterns and correlates of mental health and substance use services engagement | 12 months
  Combined analysis of mental health and substance use services engagement as measured by self report. Patterns and correlates of engagement will be measures using data from self report surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States